CLINICAL TRIAL: NCT03590665
Title: Central & Peripheral Blood Flow Regulations in Individuals With Down Syndrome
Brief Title: Blood Flow in Individuals With Down Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI accepted a position at a new Institution and terminated the study at UIC.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thessa Hilgenkamp, Postdoctoral fellow, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2017-0642; 1K99HD092606-01 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-18 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Down Syndrome
Keywords: exercise, blood flow, strength, blood pressure, heart rate,
MeSH Terms: conditions — Down Syndrome; Motor Activity | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: The acute response to exercise in blood flow is non-invasively assessed in group of individuals with Down syndrome and a control group of age- and sex-matched individuals without Down syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Down syndrome (Other): For participants with Down syndrome, the first visit includes baseline measures and familiarization with the graded maximal exercise test protocol. If necessary, additional familiarization sessions will be scheduled for people with Down syndrome. The second visit, we perform the graded maximal exercise test and familiarize the participant with the procedures for the third visit: the hand grip exercise protocol and the lower body negative pressure (LBNP) box. The third visit we assess the peripheral blood flow during the hand grip exercise protocol without and with the LBNP. For control subjects, the first and second visit are combined. Their second visit is the same as the third visit for individuals with Down syndrome.
  Interventions: Other: Hand grip exercise and lower body negative pressure
- Individuals without Down syndrome (Other): For participants with Down syndrome, the first visit includes baseline measures and familiarization with the graded maximal exercise test protocol. The second visit, we perform the graded maximal exercise test and familiarize the participant with the procedures for the third visit: the hand grip exercise protocol and the lower body negative pressure (LBNP) box. The third visit we assess the peripheral blood flow during the hand grip exercise protocol without and with the LBNP. For control subjects, the first and second visit are combined. Their second visit is the same as the third visit for individuals with Down syndrome.
  Interventions: Other: Hand grip exercise and lower body negative pressure

INTERVENTIONS:
Other: Hand grip exercise and lower body negative pressure — For participants with Down syndrome, the first visit includes baseline measures and familiarization with the graded maximal exercise test protocol. If necessary, additional familiarization sessions will be scheduled for people with Down syndrome. The second visit, we perform the graded maximal exercise test and familiarize the participant with the procedures for the third visit: the hand grip exercise protocol and the lower body negative pressure (LBNP) box. The third visit we assess the peripheral blood flow during the hand grip exercise protocol without and with the LBNP. For control subjects, the first and second visit are combined. Their second visit is the same as the third visit for individuals with Down syndrome.

SUMMARY:
This study focuses on physiological explanations of difficulties with physical activity and exercise in individuals with Down syndrome, by non-invasively examining cardiac output and the regulation of blood flow to working muscles during exercise.

DETAILED DESCRIPTION:
Work capacity is an important predictor of declining health or physical function, and of mortality, and is commonly measured as peak oxygen consumption. Peak oxygen consumption is very low in individuals with Down syndrome, the most prevalent genetic cause of intellectual disability. Previous research suggests individuals with Down syndrome may experience a double disadvantage when they are exercising: they may not be able to increase cardiac output sufficiently and they may not be able to allocate adequate blood flow to the working muscles.

The aim of this research study is therefore to determine the impact of limitations in central and peripheral regulation of blood flow on work capacity in individuals with DS. The results of this project will aid our understanding of the underlying mechanisms and determine the potential to improve health across the lifespan of individuals with Down syndrome by tailoring exercise interventions.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years old
* generally healthy
* sedentary or low-active (defined as being involved in less than 30 minutes of moderately-intense physical activity per day)
* additionally for the participants with Down syndrome:

  * diagnosis of Down syndrome trisomy 21 and
  * normal thyroid function or stable thyroid function (and medications) for at least 6 months.

Exclusion Criteria:

* atherosclerotic or other vascular disease;
* asthma or other pulmonary disease;
* hypertension (defined BP >140/90 mmHg);
* blood pressure below 90/60 mmHg;
* history of pre-syncope or syncope;
* diabetes (defined as Hba1c of >7.5% or use of glucose lowering medication);
* severe obesity (defined as BMI >40);
* medications affecting heart rate, blood pressure or arterial function;
* anti-inflammatory medication including NSAIDS;
* current smoking and
* pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Brachial blood flow | In minute 4 of the 5-minute bout of grip strength exercise
  Forearm blood flow and vascular conductance will be measured in both the exercising and non-exercising arm using high definition ultrasound (Alpha 7, Aloka-Hitachi). The brachial artery will be imaged in dual mode allowing for simultaneous determination of artery diameter (B-mode) and flow velocity (Doppler mode). Blood flow will be determined from the following formula: Forearm Blood flow = (Mean blood velocity) x (Brachial Cross Sectional Area) x (60) and expressed as ml/min. Forearm vascular conductance will be determined by dividing forearm blood flow by mean arterial pressure. Forearm blood flow and vascular conductance will be normalized to forearm lean mass to account for differences in lean mass between individuals.

SECONDARY OUTCOMES:
Muscle oxygenation | In minute 4 of the 5-minute bout of grip strength exercise
  Muscle oxygenation will be measured with near-infrared spectography (NIRS), which is a simple, noninvasive method for measuring the presence of oxygen in muscle. It can monitor changes in muscle oxygenation and blood flow during submaximal and maximal exercise. During exercise, the extent to which skeletal muscles deoxygenate varies according to the type of muscle, type of exercise and blood flow response.
Cardiac outut | Every second minute until the 12th minute of the maximal test.
  Cardiac output will be measured during a graded maximal test protocol using ultrasonography, by measuring the aortic diameter at the level of the valve form the peristernal long axis. Ascending aortic blood flow will be measured using continuous Doppler echocardiography using a pedoff probe in the suprasternal notch.

CONTACTS AND LOCATIONS:
Overall Officials: Thessa Hilgenkamp, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Disability, Health, and Social Policy Building, Integrative Physiology Laboratory, Suite 158 at 1640 W. Roosevelt Rd, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No